CLINICAL TRIAL: NCT00750087
Title: Non-interventional Study to Observe Treatment Efficacy in Maintaining Symptoms Control in Patients With Schizophrenia, Treated With Seroquel XR
Brief Title: Non-interventional Study -Observe Treatment Efficacy in Maintaining Symptoms Control in Schizophrenia With Seroquel XR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans Eriksson - Medical Science Director, AstraZeenca
Other Study IDs: NIS-NRO-SER-2008/1
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Schizophrenia patients stabilized on Seroquel XR

SUMMARY:
the primary purpose of the study is to observe symptoms control in schizophrenia for 6 months in patients treated with Seroquel XR.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have a diagnosis of schizophrenia , as defined by DSM-IV-TR and their symptoms are controlled with Seroquel XR therapy started approximately 1 month before
* All eligible patients will be included in the protocol provided they will receive detailed information in advance and will sign consent to grant access to their own data collected during this programme.

Exclusion Criteria:

* All the patients who have a known hypersensitivity to Seroquel XR/quetiapine or any of its excipients will not be included in this study.
* As per valid Romanian SmPC, concomitant medication, that could result in drug interactions and could jeopardise patient safety will be carefully considered before having the patient enrolled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The programme will include schizophrenia patients stabilized on Seroquel XR from community sample
Sampling Method: Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale - BPRS | monthly/ at every clinic visit- 7 times

SECONDARY OUTCOMES:
Clinical Global Impression Severity of Illness - CGI -S | monthly/ at every clinic visit- 7 times
Clinical Global Impression Improvement CGI -I | monthly/ at every clinic visit except first visit- 6 times
Quality of Life Enjoyment & Satisfaction Questionnaire - Short Form ( Q - LES - Q - SF) | twice/first and last clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Costea, Study Chair — AstraZeneca
Locations (32):
- Romania (32):
  - Research Site, Alba
  - Research Site, Arad
  - Research Site, Bacau
  - Research Site, Baia Mare
  - Research Site, Bistriţa
  - Research Site, Botoșani
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Câmpina
  - Research Site, Călăraşi
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Deva
  - Research Site, Galati
  - Research Site, Giurgiu
  - Research Site, Horezu
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Ploieşti
  - Research Site, Râmnicu Vâlcea
  - Research Site, Satu Mare
  - Research Site, Sibiu
  - Research Site, Siret
  - Research Site, Slatina
  - Research Site, Slobozia
  - Research Site, Târgovişte
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
  - Research Site, Zalău